CLINICAL TRIAL: NCT03089502
Title: A Randomized Control Trial of the Efficacy of a Cardio-Oncology Rehabilitation Exercise Program to Improve Cardiorespiratory Fitness in Women With Breast Cancer and Treatment Related Cardiotoxicity (CORE Study).
Brief Title: Efficacy of Cardio-Oncology Rehabilitation Exercise for Women With Breast Cancer and Treatment Related Cardiotoxicity
Acronym: CORE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited recruitment
Sponsor: University Health Network, Toronto (Other)
Collaborators: MSH-UHN AMO Innovation Fund (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CORE
Record Dates: First submitted 2017-03-16; First posted 2017-03-24 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer; Left Ventricular Dysfunction; Heart Failure, Systolic
Keywords: Exercise; Cardiac Rehabilitation; Breast Caner; Left Ventricular Dysfunction; Trastuzumab; Anthracyclines
MeSH Terms: conditions — Breast Neoplasms; Ventricular Dysfunction, Left; Heart Failure, Systolic; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Rehabilitation (Experimental): The intervention group will participate in the exercise rehabilitation program for a total of 12 weeks. This includes performing aerobic training five times per week and resistance training two to three times per week. Participants will also be expected to attend the education sessions following their supervised exercise rehabilitation sessions each week.
  Interventions: Other: Exercise Rehabilitation
- Usual Care (No Intervention): Participants in the control group will be encouraged to continue with their regular physical activity routine and will receive regular standard of care by their Cardiologist and Oncologist.

INTERVENTIONS:
Other: Exercise Rehabilitation — The intervention will consist of a walking or biking program performed at an intensity of 60-80% of VO2peak, progressing to a minimum of 150 minutes/week. Each session will include a warm up and cool down. One weekly exercise session will be supervised and participants will be expected to complete four additional aerobic training sessions at home or in the community each week. Resistance training will be introduced during the 4th week of the program and will consist of 10 exercises targeting all major muscle groups. One weekly resistance training session will be supervised following the aerobic training, and participants will be expected to complete one to two additional sessions at home or in the community each week. Weekly education sessions will follow the supervised exercise session.
  Arms: Exercise Rehabilitation

SUMMARY:
Breast cancer is the leading cause of cancer among Canadian women with nearly 26,000 new cases diagnosed each year. Fortunately, advancements in diagnostic tools and curative treatments have significantly improved overall survival. However, the development of cardiac toxicity (including asymptomatic and symptomatic heart failure) associated with use of anthracycline containing chemotherapy and targeted therapies including trastuzumab limits improvements in survival for women with breast cancer. Cardiac toxicity is a life threatening complication that leads to reduced physical functioning and quality of life. The increased risk is associated with shared risk factors among cancer and heart failure and the direct influence of cancer therapy on the cardiovascular system. Cardiac rehabilitation (CR) (including exercise training and education/counselling) has been shown to improve health outcomes, reduce heart failure related hospitalizations and modestly improve mortality among individuals with non-treatment related heart failure and may benefit women with breast cancer and treatment related cardiac toxicity (BC-CT). Therefore, this single centre, randomized control trial aims to determine if participation in an exercise based CR program can improve cardiorespiratory fitness, cardiovascular function/structure and health, and quality of life among women with BC-CT.

DETAILED DESCRIPTION:
Study Design: A single centre, two-arm, parallel group with standard of care controlled superiority trial with a balanced (1:1) block randomization will be conducted at the Toronto Rehabilitation institute, Toronto Canada. A total of 38 women (19 participants per study arm) with BC-CT presenting at Cardiology Clinics in Toronto Canada will be enrolled. After baseline assessments, eligible participants will be randomized to one of two arms including the exercise rehabilitation program or the control group (no exercise training intervention).

Patient Population: Women with BC-CT (defined as a decrease in the left ventricular ejection fraction of >10 percentage points, to a value <53% by 2D-echocardiography or a diagnosis of heart failure) who are undergoing therapy with anthracyclines and/or trastuzumab.

Procedures: The following measurements will be collected at the beginning and following the 12 week intervention. Participants will also be expected to attend one weekly exercise session at the Toronto Rehabilitation institute each week, and will be expected to complete additional exercise training sessions at home or in the community each week.

Day 1: All participants will then undergo baseline assessments at the Toronto Rehabilitation Institute including a cardiopulmonary exercise test to assess VO2peak. Resting and exercise haemodynamic outcomes, VO2peak achieved, symptoms, and reason for test termination will also be collected. Standard measures conducted during the intake process including height, weight, body fat percent, and waist circumference will also be collected. The participants will be provided with a blood requisition form that will be returned during the first week of class. The questionnaires for physical activity patterns (Godin Leisure Physical Activity Questionnaire), quality of life, a health history questionnaire, as well as the activity tracking devices will also be administered by the research coordinator upon their initial visit.

Day 2: All cardiac assessments will be conducted on a separate day of testing at Toronto General Hospital by a skilled clinical cardiac sonographer.

Day3: The vascular assessment will be completed at the University of Toronto.Trained research staff familiar with echocardiography analysis will complete all offline analyses for the vascular assessments.

Throughout the program: Information regarding adherence to the exercise program will also be collected by the research coordinator each week via the exercise training diaries and activity tracking devices from each participant. Reasons for missed sessions will also be assessed. Lastly, completion rates of the program will be collected via the patient chart upon completion of their final cardiopulmonary exercise test.

Intervention: The exercise rehabilitation program will consist of one weekly supervised 90-minute session consisting of aerobic and resistance exercise in addition to education/counselling for a total of 12 weeks. Each participant will be asked to complete four additional aerobic training sessions and one to two resistance training sessions at home or in the community each week. Case managers including nurses, physiotherapists and registered kinesiologists will be responsible for supervising each class. The participants initial aerobic exercise prescription will be based on outcomes from the baseline cardiopulmonary exercise test. The first week of class will include an initial exercise trial to determine if the exercise prescription based on the cardiopulmonary exercise test is appropriate for the individual (i.e., similar heart rate response to exercise, the participant can complete the exercise prescription and any potential symptoms that might be reported). Participants will engage in over-ground walking, treadmill walking or stationary biking depending on the limitations of the individual, participant preference and availability of equipment to complete the exercise at home. The goal is to progress patients to 60 minutes of aerobic exercise, five times per week, at intensity equivalent to 60% to 80% of VO2peak, which is equivalent to an intensity that is just below the ventilatory threshold. Exercise duration will be increased every one to two weeks (equivalent to 10% of the current exercise prescription duration), with a maximum intensity of 80% of VO2peak. The exercise prescription will be progressed based on feedback from the patient, exercise heart rate and rating of perceived exertion. Participants will be able to monitor the exercise prescription using the heart rate achieved on the cardiopulmonary exercise test that corresponds to 60% to 80% of VO2peak and a rating of perceived exertion that corresponds to 11 to 15 on the Borg scale. Patients will be required to keep a detailed record of each exercise session, noting distance walked/biked, duration, resting and peak heart rate, and rating of perceived exertion for each aerobic training session.

Resistance training will be introduced during the 4th week of the program. The resistance exercise program will consist of ten exercises targeting all major muscle groups. Participants will begin with 10 repetitions at a weight that is equivalent to 60 to 70% of the individuals 1 repetition maximum. The weight required to achieve this exercise intensity will be determined in the 4th week of class using a modified 1 repetition maximum assessment. The resistance training will then be progressed every 1 to 2 weeks increasing the number of repetitions to 12 and 15 respectively. Once the participant can complete 15 repetitions, they will be instructed to reduce the repetitions back to 10 and add an additional set. The same progression will be used until the participants can complete 3 sets of 15 repetitions. Resistance training records will include the amount of weight lifted, the number of repetitions completed, sets performed and rating of perceived exertion during each exercise.

Education Component: Each week participants will attend a 30-minute education session following completion of their exercise training. The education component of the program will consist of topics that are designed to help participants achieve optimal self-management of their conditions and foster lifestyle behavior change. The education sessions delivered will be consistent with the current education program at the Toronto Rehabilitation Institute. Topics that will be addressed in the educational sessions will include, but are not limited to, the benefits of physical activity, goal setting, healthy eating, dealing with stress and coping, and management of the toxic effects of treatments for breast cancer. Qualified staff including kinesiologists, physiotherapists, dietitians and psychologists will deliver the education sessions.

Control Group (No Exercise Intervention): Participants who are randomized the control group will undergo baseline and follow up assessments at 12 weeks. They will not have any other contact with the study staff over the duration of the study period. They will also be asked to continue with their regular physical activity routine and will be medically managed as per standard of care by their Cardiologist and Oncologists. All participants will also complete the Godin Leisure Time Physical Activity Questionnaire to determine if there are potential increases in physical activity in the exercise and control group, which may account for changes in all outcome measures. All participants in each group will also be asked to wear an activity-tracking device, including a step counter (PiezoRx®) for one week before and following the intervention (12 weeks) to objectively quantify their daily physical activity. After program completion the control group participants will be provided with the opportunity to enroll in the exercise-rehabilitation program in order to have the opportunity to benefit from the program.

Timeline of Trial: The target of this trial is to demonstrate superiority. The trial will last a total of 12 weeks. All outcomes (primary and secondary) will be measured at baseline and following the intervention.

Randomization: Randomization will occur at the central site, the Toronto Rehabilitation Institute, using a computer generated randomization schedule with an allocation ratio of 1:1.

Blinding: The participants will not be blinded to their intervention arm. Assessors of outcome data and analysis will be blinded to the intervention arm.

Analytical Plan: The principal analysis of the primary outcome will employ an intention-to-treat analysis and will include all randomized participants in their randomly assigned group. The primary and secondary analyses will include continuous variables with baseline differences between the two groups to be analyzed using a one way-analysis of variance. Continuous variable outcomes with values over the two time periods will be analyzed using a repeated measures analysis of covariance, with the baseline values treated as covariates. A multiple regression model will also be used to compare study arms relative to the change in physiological mediators (e.g. cardiac function and vascular endothelial function) of the aerobic training to the change in VO2peak relationship. These analyses will be conducted to determine whether physiological variables mediate the effect of exercise training on VO2peak. Finally, two separate regression models will used to address how changes in VO2peak will affect changes in quality of life using the two separate measures (model A and model B) following completion of the program.

Significance: Outcomes of this investigation will provide insight for potential therapeutic interventions to improve adverse events associated with treatments for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer (receptor status: human epidermal growth factor receptor (HER2+/-), Progesterone receptor, (PR+/-), estrogen receptor (ER+/-); Stage I-III)
* Are 18 yrs. of age or older
* A diagnosis of cardiac toxicity that occurred during treatment will be defined as a decrease from baseline in the left ventricular ejection fraction of >10 percentage points, to a value < 53% by 2D-echocardiography upon repeated measures or a diagnosis of heart failure which will be confirmed by the cardiologist upon cardiac evaluation
* Currently undergoing known cardiotoxic agents including the HER2-antagonist trastuzumab and/or chemotherapy agents including doxorubicin and epirubicin

Exclusion Criteria:

* Women who are pregnant
* Treated with a left ventricular assistant device or a pacemaker.
* Have metastatic disease
* Previous exposure to anthracyclines, cytotoxic treatments or radiation preceding their breast cancer diagnosis
* Unable to confirm a diagnosis of heart failure due to treatment for breast cancer upon cardiac evaluation by their Cardiologist
* Myocardial infarction, complex arrhythmias, or unstable cardiac symptoms in the previous six weeks prior to study enrolment
* Significant co-morbidities that limit their ability to perform exercise (i.e., severe peripheral artery disease, severe chronic obstructive pulmonary disease, musculoskeletal injury or stroke)
* Contraindications to exercise training identified on their first cardiopulmonary assessment that do not subside prior to beginning the program including angina pectoris symptoms, light-headedness or dizziness with exercise, and resting blood pressure > 200mmHg systolic or >120mmHg diastolic blood pressure.
* Contraindications to resistance training including increased eye pressures (> 20mmHg), untreated hernias, limitations due to surgery (lumpectomy/mastectomy) and potential musculoskeletal injuries

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Fitness | Baseline and 12 weeks
  A cardiopulmonary exercise test will be completed following the Bruce or modified Bruce protocol. Breath-by-breath gas samples will be collected and averaged over a 20-second period using a calibrated metabolic cart (Vmax Encore, SensorMedics, Yoba Linda, CA).

SECONDARY OUTCOMES:
Cardiovascular Risk Profile | Baseline and 12 weeks
  This will be assessed using a standard blood requisition blood form including measurement of lipids, cholesterol, and triglyceride levels. Anthropometrics including body mass index, waist circumference, body fat percent and hemodynamic profiles including heart rate, systolic and diastolic blood pressure values (resting and during exercise) will also be collected.
Cardiac Function and Structure at Rest | Baseline and 12 weeks.
  2D Echocardiography will be used for the measurement of left ventricular volumes, cardiac output, stroke volume, left ventricular ejection fraction, diastolic function, left ventricular wall thickness and left ventricular cavity size. Strain and Strain Rate via 2D-Speckle tracking imaging will also be collected at rest to assess cardiac function.
Cardiac Function During Stress (Exercise) | Baseline and 12 weeks
  Exercise will be performed following a standardized stress echocardiography protocol. 2D-echocardiography assessments will be conducted at rest, during exercise and within 30 seconds of exercise completion.
Endothelial Function | Baseline and 12 weeks
  Endothelial dependant flow mediated dilation of the brachial artery will be assessed using a portable ultrasound unit (Vivid 9E GE Healthcare), and a 8-14-MHz transducer (GE Medical Systems Wauwatosa, WI USA).
Arterial Stiffness | Baseline and 12 weeks
  Arterial Stiffness will be measured by pulse-wave velocity (Sphygmocor® system).
Autonomic Function | Baseline and 12 weeks
  Baroreceptor sensitivity will be collected as a measure of autonomic function. Each participant will be secured with a three-lead ECG and finger plethysmography worn on the middle finger, while measures of a beat-by-beat blood pressure are recorded (Finapres; Ohmeda Inc, Englewood, CO).
Quality of Life | Baseline and 12 weeks
  The Kansas City Cardiomyopathy Questionnaire will be used to assess health related quality of life for heart failure.
  The FACT-B questionnaire will be used as a measurement of health related quality of life for individuals with breast cancer.

OTHER OUTCOMES:
Exercise Adherence | Throughout the exercise training program (up to 12 weeks)
  Adherence will be assessed using an attendance sheet for each the supervised sessions. If participants do not complete their target exercise prescription, the reasons will be recorded. The participants will also complete weekly exercise diaries at home each week and will be asked to record reasons for missed sessions or if they were unable to meet their exercise prescription. A step counter (PiezoRx®) that monitors the participants' moderate/vigorous activity time (>100 steps per minute) as well as bouts per week (greater than 10 minutes of moderate/vigorous activity) will also be recorded. These measurements will be used to confirm the reported exercise sessions to be completed at home each week.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Oh, MD,MSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual data of the primary and secondary outcomes will be made available to other researchers as a supplementary file to be accompanied by any publications generated by this clinical trial. Individual data will also be made available upon request for research purposes